CLINICAL TRIAL: NCT01996202
Title: A Pilot Study of Ipilumimab and Radiation in Poor Prognosis Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00045042
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: High Risk Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resected Melanoma (Other): Subjects with resected melanoma.
  Interventions: Drug: Ipilumimab; Radiation: Radiation
- Unresected Melanoma (Other): Subjects with unresected melanoma.
  Interventions: Drug: Ipilumimab; Radiation: Radiation

INTERVENTIONS:
Drug: Ipilumimab
Radiation: Radiation

SUMMARY:
This is a pilot study assessing the safety of the combination of ipilimumab administered concurrently with radiotherapy for patients with locally advanced or unresectable melanoma and patients at high risk for recurrence after resection.

ELIGIBILITY:
Inclusion criteria:

1. Willing and able to give written informed consent.
2. Histologic diagnosis of melanoma
3. Cohort 1: Resected patients at high risk of recurrence. Patients must meet at least one of the following criteria

   a. Melanoma of mucosal origin b. Desmoplastic melanoma c. Primary melanoma of the head or neck with any lymph node involvement d. Patients with non-head and neck primaries must have had preoperative/pathologic macroscopic lymph node involvement, defined by clinically evident on exam or imaging evaluation, plus at least one of the following by clinical, imaging, or pathologic evaluation: i. ≥ 2 cervical or axillary nodes ii. ≥ 3 groin lymph nodes iii. Extracapsular extension (ECE) of tumor iv. Lymph nodes ≥ 3cm
4. Cohort 2: Neoadjuvant/definitive approach for locally advanced patients. Patients must meet at least one of the following criteria

   1. Melanoma of mucosal origin
   2. Desmoplastic melanoma
   3. Patients with radiographic evidence of tumor invasion into surrounding local structures rendering them inoperable
   4. Macroscopic nodal involvement. In addition, patients must also meet one of the following criteria

   i. Recurrent disease, with any number and size of nodes ii. ≥ 1 parotid node(s) iii. ≥ 2 cervical or axillary nodes iv. ≥ 3 groin lymph nodes v. Lymph nodes ≥ 3cm vi. ECE of tumor
5. Resected patients should begin treatment within 12 weeks of surgery, once adequately healed as determined by the treating physicians.
6. Local-regional treatment sites must be able to be encompassed within a reasonable radiation therapy treatment volume
7. Patients with recurrent disease are allowed in cohort 1, provided at least one of the criteria listed in 3 above is met
8. For patients with a new diagnosis of melanoma treated in cohort 2 who have a cutaneous primary, the primary site may be addressed surgically (wide local excision; skin grafting) prior to the initiation of ipilimumab and radiation at the discretion of the treating surgeon.
9. Required values for initial laboratory tests:

   * WBC ≥ 2000/uL
   * ANC ≥ 1000/uL
   * Platelets ≥ 75 x 103/uL
   * Hemoglobin ≥ 9 g/dL (≥ 80 g/L; may be transfused)
   * Creatinine ≤ 2.0 x ULN
   * AST/ALT ≤ 2.5 x ULN
   * Bilirubin ≤ 2.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
10. No active or chronic infection with HIV, Hepatitis B, or Hepatitis C.
11. ECOG performance status ≤ 1
12. Men and women, ≥ 18 years of age
13. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized

    WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as:
    * Amenorrhea ≥ 12 consecutive months without another cause, or
    * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level ≥ 35 mIU/mL.

    Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.

    WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours before the start of ipilimumab.

    Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and for up to 26 weeks after the last dose of investigational product] in such a manner that the risk of pregnancy is minimized.
14. Patients must agree to blood sampling to participate in study.

Exclusion criteria:

1. Ocular melanoma
2. Presence of brain metastases
3. Prior radiation therapy for melanoma
4. Any other malignancy form which the patient has been disease-free for less than 3 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix, or DCIS. Patients with prior malignancies that are not considered to be an active problem may be enrolled at the discretion of the investigator, regardless of time frame.
5. Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).
6. Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
7. Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
8. A history of prior treatment with ipilimumab or prior CD137 agonist or CTLA 4 inhibitor or agonist.
9. Concomitant therapy with any of the following: IL 2, interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids in the previous 4 weeks (defined as prednisone 10mg daily or equivalent.)
10. Women of childbearing potential (WOCBP), defined above in Section 4.1, who:

    1. are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 26 weeks after cessation of study drug, or
    2. have a positive pregnancy test at baseline, or
    3. are pregnant or breastfeeding.
11. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness.
12. Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 26 weeks after ipilimumab is stopped. Sexually active WOCBP must use an effective method of birth control during the course of the study, in a manner such that risk of failure is minimized. Before study enrollment, WOCBP must be advised of the importance of avoiding pregnancy during study participation and the potential risk factors for an unintentional pregnancy. All WOCBP MUST have a negative pregnancy test before first receiving ipilimumab. If the pregnancy test is positive, the patient must not receive ipilimumab and must not be enrolled in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Incidence of immune related adverse events associated with ipilimumab | 2 years
Incidence of acute and late radiation toxicities | 2 years

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 years
6 month progression free survival (PFS) | 6 months
12 month progression free survival (PFS) | 12 months
Overall survival | 2 years
CD4+ and CD8+ reactivity to melanoma tumor antigens | 2 years
Cytokines associated with anti-tumor response | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States